CLINICAL TRIAL: NCT02147977
Title: Effects of Marine n-3 Fatty Acids on Heart Rate Variability and Arrhythmias in Patients Receiving Chronic Dialysis (Renal Rhythm Study II)
Brief Title: Effects of Marine n-3 Fatty Acids on Heart Rate Variability and Arrhythmias in Patients Receiving Chronic Dialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Jesper Moesgaard Rantanen, MD, Aalborg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: N-20140013
Record Dates: First submitted 2014-05-21; First posted 2014-05-28 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Kidney Failure Chronic; Arrhythmias Cardiac
Keywords: Renal Dialysis; Arrhythmias Cardiac; Death Sudden Cardiac; Fatty Acids Omega 3
MeSH Terms: conditions — Renal Insufficiency, Chronic; Arrhythmias, Cardiac; Death, Sudden, Cardiac | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dietary supplement: n-3 PUFA (Active Comparator): n-3 polyunsaturated fatty acids from fish oil
  capsules of 500 mg. 2 g a day.
  Interventions: Dietary Supplement: dietary supplement: n-3 PUFA
- olive oil (Placebo Comparator): Capsules of 500 mg. 2 g a day.
  Interventions: Dietary Supplement: olive oil

INTERVENTIONS:
Dietary Supplement: dietary supplement: n-3 PUFA
  Other Names: Calamarine 250/250 TG
  Arms: dietary supplement: n-3 PUFA
Dietary Supplement: olive oil
  Arms: olive oil

SUMMARY:
Background: End Stage Renal Disease (ESRD) patients have an extremely high mortality and the leading cause of death is cardiovascular disease which accounts for 50% of all deaths. It is estimated that about one third is due to arrhythmias. Previous studies reveal a higher risk of various arrhythmias in dialysis patients but the prevalence is uncertain. Atrial fibrillation is the most common arrhythmia among patients with ESRD. The arrhythmia is often asymptomatic, but the risk of stroke increases dramatically and the annual mortality doubles. Autonomic cardiac dysfunction is often seen in patients with ESRD, and this is expressed by attenuated Heart Rate Variability (HRV) which is a measure of the variation in the time interval between heart beats. Attenuated 24 hours HRV is associated with an increased risk of sudden cardiac death in the general population and among patients with ESRD. N-3 polyunsaturated fatty acids (PUFAs) in fish or fish oil supplements have been shown to increase HRV and reduce the risk of various ventricular and supraventricular arrhythmias in some but not all studies, but this effect has only been sparsely investigated in the high risk patients with ESRD, who has a very low intake of n-3 PUFAs.

Objective: The purpose of this study is to investigate the effects of n-3 PUFA supplementation on HRV and arrhythmias in dialysis patients.

Hypothesis: n-3 PUFA supplementation increases 24 hours HRV in dialysis patients. n-3 PUFA supplementation reduces the level of Supraventricular tachycardia, premature atrial complexes (PACs) and premature ventricular complexes (PVCs) in chronic dialysis patients.

Design: Randomized double-blind, placebo controlled trial

Study participants: 140 dialysis patients at Aalborg University Hospital and Vendsyssel Hospital, Hjørring in Denmark.

Inclusion time: Summer 2014 to Fall 2015

Methods: The patients are allocated to 3 months treatment with supplements of 2 g n-3 PUFAs or placebo (olive oil). The following data are registered at baseline and after 3 months treatment: Demographics and medical history, Standard ECG-12, blood pressure, blood samples, 48 hours ambulatory ECG Holter recordings, Intake of n-3 PUFAs (assessed by questionnaires and blood measurements).

Perspective: A positive result of this study might make it possible to achieve a reduction in arrhythmias and mortality in these high risk patients by a cheap and well tolerated nutritional supplement.

ELIGIBILITY:
Inclusion Criteria:

* Dialysis > 3 months
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* Patients who is not able to consent.
* Known allergy to contents of the olive or fish oil capsules.
* Remaining life expectancy < 3 months.
* Pregnancy (positive S-HCG) - test only performed in cases of doubt.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2014-06; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in the 24 hours time domain index: standard deviation of NN-intervals (SDNN) in milliseconds (ms) | baseline and 3 months
  Evaluated using 48 hours Holter ECG recordings at baseline and after 3 months.

SECONDARY OUTCOMES:
change in number of episodes with supraventricular tachycardia per day | baseline and 3 months
  evaluated using 48 hours Holter ECG recordings at baseline and after 3 months.
change in number of premature atrial complexes per day | baseline and 3 months
  evaluated using 48 hours Holter ECG recordings at baseline and after 3 months.
change in Lown class of premature ventricular complexes | baseline and 3 months
  Evaluated using 48 hours Holter ECG recordings at baseline and after 3 months.

OTHER OUTCOMES:
change in frequency domain indices of heart rate variability | baseline and 3 months
  total power (TP), Ultra low frequency (ULF), Very low frequency (VLF), low frequency (LF), high frequency (HF) and LF/HF.
  Evaluated using 48 hour Holter ECG recordings at baseline and after 3 months
change in other 24 hour time domain indices of heart rate variability | baseline and 3 months
  mean NN (ms), sNN50 (counts), sNN6%(counts), SDNNi (ms), SDANN (ms), RMSSD (ms), triangle index.
  Evaluated using 48 hours Holter ECG recordings at baseline and after 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper M Rantanen, MD, Principal Investigator — Department of Nephrology Aalborg University Hospital; Jeppe H Christensen, DMSc, Study Director — Department of Nephrology Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Department of Nephrology, Aalborg, Denmark